CLINICAL TRIAL: NCT00158132
Title: A Double-Blind, Placebo Controlled Trial of Propranolol and Amantadine for the Treatment of Cocaine Dependent Subjects With Severe Cocaine Withdrawal Symptoms
Brief Title: Effectiveness of Amantadine and Propranolol for Treating Cocaine Dependence - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Dr. Kyle Kampman, Treatment Research Center, University of Pennsylvania
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-12756-2; P50DA012756-02 (NIH); DPMC (Other: NIDA); NCT00128349 (obsolete NCT alias)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Propranolol; Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Propranolol (Experimental): Propranolol 100mg/day in 3 divided doses
  Interventions: Drug: Propranolol
- Amantadine (Experimental): Amantadine 100mg three times daily
  Interventions: Drug: Amantadine
- Propranolol and Amantadine (Experimental): Propranolol 100mg/day in 3 divided doses and Amantadine 100mg 3X's daily
  Interventions: Drug: Propranolol; Drug: Amantadine
- Placebo (Placebo Comparator): Identical Placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol 100mg/day in 3 divided doses
  Arms: Propranolol; Propranolol and Amantadine
Drug: Amantadine — Amantadine 100mg three times daily
  Arms: Amantadine; Propranolol and Amantadine
Drug: Placebo — Placebo pills
  Arms: Placebo

SUMMARY:
Cocaine addiction is a serious health problem with no available medical treatment for preventing relapse. Amantadine, a medication that improves muscle control, and propranolol, a medication that lowers blood pressure, may be useful in treating cocaine addiction in individuals with severe cocaine withdrawal symptoms. This study will evaluate the effectiveness of amantadine and propranolol in preventing drug relapse among cocaine addicts.

DETAILED DESCRIPTION:
Cocaine withdrawal symptoms are a major contributing factor for why outpatient cocaine dependence treatment programs often fail. Individuals with severe cocaine withdrawal symptoms often experience anxiety, shaking, and muscle pain. Amantadine is a medication currently used to improve muscle control, reduce shaking, and lessen stiffness. Therefore, it may help reduce the muscle pain that some cocaine addicts experience. By enhancing activity of the brain chemical dopamine, amantadine may also reduce other symptoms associated with cocaine withdrawal. Propranolol is a medication currently used to treat high blood pressure and irregular heart rhythms. It may reduce anxiety and lessen cocaine cravings in individuals addicted to cocaine. The purpose of this study is to evaluate the effectiveness of amantadine and propranolol, alone and in combination, for treating cocaine addicts with severe cocaine withdrawal symptoms.

A 2-week baseline evaluation period will be followed by an 8-week treatment phase. During the baseline evaluation, cocaine use will be measured with urine tests, three times each week. Only participants who are experiencing severe withdrawal symptoms and who use cocaine at least twice during the first 2 weeks will continue in the study. Eligible individuals will then be randomly assigned to receive amantadine alone, propranolol alone, a combination of amantadine and propranolol, or placebo. Treatments will begin at Week 3 and study visits will occur three times each week. Cocaine levels will be monitored throughout the study with urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, 18 to 60 years old.
* Meets DSM-IV diagnosis criteria for cocaine dependence as determined by the Structured Clinical Interview for DSM-IV (SCID)
* Score of at least (> or =) 22 on the Initial Cocaine Selective Severity Assessment (CSSA)
* Lives within commuting distance of the Treatment Research Center (TRC) and the Penn/VA Center for Studies of Addiction, University of Pennsylvania
* If female, willing to use contraception throughout the study
* Continued use of cocaine during a two week evaluation phase prior to medication treatment as demonstrated by at least 2 new uses of cocaine documented by quantitative urine toxicology screen obtained three times weekly according to new use rules

Exclusion Criteria:

* Meets DSM-IV/SCID diagnosis criteria for dependence on any drugs other than cocaine, marijuana, or nicotine. Cocaine dependent subjects who identify cocaine dependence as their primary addiction but who also meet criteria for alcohol dependence will be accepted as long as the alcohol dependence is not severe enough to require medications for alcohol detoxification.
* Concomitant treatment with psychotropic medications.
* Patients mandated to treatment based upon a legal decision or as a condition of employment. This will be assessed by the patient's self-report.
* Current severe psychiatric symptoms (e.g., psychosis, dementia, suicidal or homicidal ideation, mania or depression requiring antidepressant medication)
* Sensitivity to propranolol or amantadine
* Use of any investigational medication within the past 30 days.
* History of significant heart disease (an arrhythmia which required medication, Wolff-Parkinson -White Syndrome, angina pectoris, documented history of myocardial infarction, heart failure).
* History of chest pain associated with cocaine use which has prompted a visit to a physician.
* Current use of reserpine, verapamil, theophylline, trimethoprim, cimetidine, haloperidol, benzodiazepines, or anticonvulsants
* Bronchospastic disease
* Hyperthyroidism
* Diabetes mellitus
* Patients with known AIDS or other serious illnesses which may require hospitalization during the study.
* Female subjects who are pregnant or lactating, or female subjects of child bearing potential who are not using acceptable methods of birth control. Acceptable methods of birth control include:

  1. barrier (diaphragm or condom) with spermicide
  2. intrauterine progesterone contraceptive system
  3. levonorgestrel implant
  4. medroxyprogesterone acetate contraceptive injection
  5. oral contraceptives.
* Patients with impaired renal function as indicated by corrected creatinine clearance below 80 ml/min/70 kg as determined by the modified Cockcroft equation (CDC, 1986).
* Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the Principal Investigator. EKG 1st degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed; liver function tests [LFTs] <5 x ULN are acceptable). A complete list of exclusionary lab results are included in the appendix 1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 1999-09; Primary Completion 2005-03 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Cocaine abstinence; measured by self-reported Time line follow-back and confirmed with cocaine urine tests. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helen M. Pettinati, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Kampman KM, Dackis C, Lynch KG, Pettinati H, Tirado C, Gariti P, Sparkman T, Atzram M, O'Brien CP. A double-blind, placebo-controlled trial of amantadine, propranolol, and their combination for the treatment of cocaine dependence in patients with severe cocaine withdrawal symptoms. Drug Alcohol Depend. 2006 Nov 8;85(2):129-37. doi: 10.1016/j.drugalcdep.2006.04.002. Epub 2006 May 11. PMID 16697124
- See also: Related Info — http://www.med.upenn.edu/csa/index.html